CLINICAL TRIAL: NCT02334202
Title: Preventing Obesity in Military Communities, Adolescents (POMC-Adolescents)
Brief Title: Preventing Obesity in Military Communities, Adolescents
Acronym: POMC-A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: Fort Belvoir Community Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Marian Tanofsky-Kraff, Associate Professor, Uniformed Services University of the Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F172NC-S2
Record Dates: First submitted 2014-12-23; First posted 2015-01-08 (Estimated); Last update posted 2018-08-03 (Actual); Status verified 2018-08

CONDITIONS: Obesity; Weight Gain; Disordered Eating; Eating Disorder
Keywords: Adolescent; Obesity/Psychology; Loss of Control Eating; Child; Female; Follow-Up Studies; Health Behavior; Health Education; Humans; Intervention Studies; Prospective Studies; Psychotherapy; Risk Factors; Weight Loss; Weight Gain; Military
MeSH Terms: conditions — Obesity; Weight Gain; Feeding and Eating Disorders; Health Behavior; Health Education; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health Education (Active Comparator): The health education group will follow the "HEY-Durham" health program designed by researchers at Duke University. This program, designed to be delivered to youth attending community high schools, was adapted to a 12-week program for adolescent military dependents.
  Interventions: Other: Health Education
- Interpersonal Psychotherapy-Weight Gain (Experimental): IPT-WG is designed to decrease excessive weight gain among adolescents who are at risk for adult obesity. IPT-WG involves developing strategies for dealing with the problems girls struggle with that may lead to increased eating. The IPT-WG program has been adapted to be appropriate for military dependents.
  Interventions: Behavioral: Interpersonal Psychotherapy-Weight Gain

INTERVENTIONS:
Behavioral: Interpersonal Psychotherapy-Weight Gain — Participants will have 1 individual pre-group session when each participant meets with the group leaders so that they can learn about each girl's significant relationships, set goals for the program, and so each girl can learn about group participation and format. Participants then will begin IPT-WG which is designed to decrease excessive weight gain among adolescents ages 12-17 years who are at risk for adult obesity. The IPT-WG program has been adapted to be appropriate for military dependents. The IPT-WG group meets for 12 consecutive, weekly group meetings and involves developing strategies for dealing with the problems girls struggle with that may lead to increased eating. At the 6th week of the group, the group leaders meet with each participant to review their progress and goals.
  Other Names: IPT-WG
  Arms: Interpersonal Psychotherapy-Weight Gain
Other: Health Education — The health education group will follow the "HEY-Durham" health program designed by researchers at Duke University. This program, designed to be delivered to youth attending community high schools, was adapted to a 12-week program (each with a 90 minute session). Girls will come in for a 1.5-hour group meeting once a week for 12 weeks (12 times total). Before beginning the group, girls will meet with group leaders to review each adolescent's family health history. The curriculum includes focus on various health topics, including avoiding alcohol, drug and tobacco use, nutrition and body image, nonviolent conflict resolution, sun safety, exercise, and domestic violence.
  Other Names: HEY-Durham (edited for POMC-A)
  Arms: Health Education

SUMMARY:
This research study is aimed at the prevention of excessive weight gain in female military dependents at high risk for adult obesity. The purpose of this study is to determine whether reducing Loss of Control (LOC) eating and associated indicators through use of interpersonal psychotherapy (IPT) will be feasible and acceptable to female adolescent dependents who report such behaviors. Moreover, patterns in the data will be examined to assess whether IPT influences body weight gain trajectories and prevent worsening disordered eating and metabolic functioning among female military dependents at heightened risk for unhealthy weight gain.

DETAILED DESCRIPTION:
The increased prevalence of obesity among the children of military personnel has paralleled that observed in the civilian population. Disordered eating, especially binge or loss of control (LOC) eating, is common among adolescents and is a salient risk factor for obesity and the development of exacerbated disordered eating and depressive symptoms. The goal of this study is to test the effectiveness of interpersonal psychotherapy (IPT) to slow the trajectory of weight gain in adolescent girls at high-risk for adult obesity by virtue of elevated body mass index (BMI) percentile and LOC eating. IPT targets the difficult social functioning and stressful events that are associated with LOC and highly relevant to the adolescent youth from military families. Adolescent military dependents will be randomized to receive either the IPT weight gain prevention program or a health education (HE) control condition, for 12 weekly group sessions. Adolescents' weight status, eating behaviors, and mood will be assessed at baseline, immediately following the prevention program (12-weeks), and at 1-year follow-up. At 2-year and 3-year follow-up time points, participants' BMI and physiologic data will be collected via the Military Health System's electronic medical record system. It is hypothesized that adolescents who receive the IPT group program will show significantly less weight gain (or more weight loss) relative to those randomized to HE at 3-year follow-up. Additionally, it is hypothesized that adolescents receiving IPT (as compared to HE) will demonstrate improvements on secondary outcomes of interest, including the presence and frequency of classic binge eating episodes, as well as obesity-related physiological measures of health (e.g., fasting insulin). The overall goal of the study is to prevent excess weight gain and adult obesity, and to prevent worsening disordered eating and metabolic functioning among overweight military dependents at risk for adult obesity and binge eating disorders.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Age between 12 and 17 years (at the start of the study)
* English-speaking
* Ability to complete study procedures, including ability to participate in a group
* Endorsement of at least one LOC criteria, as assessed by Eating Disorder Examination (EDE) semi structured interview

Exclusion Criteria:

* Presence of a chronic major medical illness: : renal, hepatic, gastrointestinal, endocrinologic (e.g., Cushing syndrome, hyper- or hypothyroidism), hematological problems or pulmonary disorders (other than asthma not requiring continuous medication). Non-serious medical illnesses, such as seasonal allergies, will be reviewed on a case-by-case basis.
* Presence of a documented, obesity-related medical complication that would require a more aggressive weight loss intervention approach: type 2 diabetes, hyperlipidemia, hypertension, fasting hyperglycemia, or nonalcoholic steatohepatitis
* Documented or self-reported current pregnancy, current breast-feeding, or recently pregnant girls (within 1 year of delivery). Because pregnancy is a state in which weight gain is expected and appropriate, pregnant individuals would not be suitable for this study. Sexually active females must be using an effective form of birth control. These methods include total abstinence (no sex), oral contraceptives ("the pill"), an intrauterine device (IUD), levonogestrol implants (Norplant), or medroxyprogesterone acetate injections (Depo-provera shots). If one of these cannot be used, contraceptive foam with a condom is recommended. Should a participant in the IPT-WG group become pregnant during the ~12 weeks of the group program, she will be excluded from the group sessions. The study team will closely assist in obtaining an appropriate referral to a community mental healthcare provider, as indicated, and will request a release of information so that they may facilitate a smooth transition for the girl.
* Current, regular use of prescription medications that affect appetite, mood, or body weight: currently prescribed SSRI's, neuroleptics, tricyclics, stimulants, or any other medication known to affect appetite, mood, or body weight. Oral contraceptive use will be permitted, provided the contraceptive has been used for at least two months before starting the prevention groups. Medication use for non-serious conditions (e.g., acne) will be considered on a case-by-case basis.
* Current involvement in psychotherapy or a structured weight loss program.
* Weight loss during the past two months for any reason exceeding 3% of body weight.
* Current anorexia nervosa or bulimia nervosa as determined by documented medical history or if uncovered during K-SADS semi-structured interview. Current binge eating disorder will be permitted. Girls with anorexia or bulimia nervosa will be referred to mental health specialists for further evaluation and treatment. Individuals who need further behavioral health or medical services will be accommodated through their primary care medical home in accordance with normal clinical standard of care. This will be accomplished by direct communication with the patients' primary care physician.
* Individuals who have major depressive disorder, psychoses, current substance or alcohol abuse, conduct disorder, as determined by Kiddie Schedule for Affective Disorders and Schizophrenia (K-SADS) semi-structured interview and as defined by criteria outlined in the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV-TR) or any other DSM-IV-TR psychiatric disorder that, in the opinion of the investigators, would impede competence or compliance or possibly hinder completion of the study.

Ages: 12 Years to 17 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child
Enrollment: 48 (Actual)
Dates: Start 2011-11; Primary Completion 2018-08 (Actual); Study Completion 2018-08 (Actual)

PRIMARY OUTCOMES:
Body mass index metrics | Baseline, Change from baseline at post-intervention, 1-year, and 2-year
  Participants will be weighed using professional grade equipment and trained personnel.

SECONDARY OUTCOMES:
Social and emotional functioning | Baseline, Change from baseline at post-intervention, 1-year, and 2-year
  Participant composite scores on measures of disordered eating, depressive and anxiety symptoms, as measured by an extensive battery of standardized assessments.
Blood-based metabolic markers | Baseline, Change from baseline at post-intervention, 1-year, and 2-year
  Blood drawn for measurement of triglycerides, HDL cholesterol, glucose, and other indicators of obesity risk -e.g. hormones thought to affect appetite and weight.

CONTACTS AND LOCATIONS:
Overall Officials: Marian Tanofsky-Kraff, Ph.D., Principal Investigator — Uniformed Services University of the Health Sciences
Locations (1):
- Fort Belvoir Community Hospital, Fort Belvoir, Virginia, United States

REFERENCES:
- [Background] Tanofsky-Kraff M, Sbrocco T, Theim KR, Cohen LA, Mackey ER, Stice E, Henderson JL, McCreight SJ, Bryant EJ, Stephens MB. Obesity and the US military family. Obesity (Silver Spring). 2013 Nov;21(11):2205-20. doi: 10.1002/oby.20566. Epub 2013 Sep 5. PMID 23836452